CLINICAL TRIAL: NCT01761253
Title: Assessing Costs & Cost-variability Among Enrollees of Health Insurance Programs Utilizing Charlson's Comorbidity Index and Administrative Databases
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Mary E. Charlson, MD, Executive Director, Center for Integrative Medicine/Chief, Division of Clinical Epidemiology and Evaluative Sciences Research, Weill Medical College of Cornell University
Other Study IDs: WCMC IRB No. 910010709
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Multiple Chronic Illnesses
Keywords: comorbidity, multiple chronic conditions, Medicaid, prediction of cost; Predictive models, cost containment, managed care
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Assessing costs & cost-variability: Data for the approximately 15,000 patients who were continuously enrolled during the calendar years 2006 and 2007 in the Generations Plus/ Northern Manhattan Health Network and 226,000 members of a large self insured union trust fund from 2007-2010 will be combined. The data will include age, gender, length of plan enrollment, whether or not the patient is disabled, their diagnoses, and their use of medical and social services.

SUMMARY:
This study will involve the evaluation of the cost profile of about approximately 241,000 patients (15,000 who are members of the Generations Plus/ Northern Manhattan Health Network AND 226,000 members of a large self insured union trust fund). We will test the hypothesis that as comorbidity scores exceed three-four, patients will have an exponential increase in average yearly cost with a parallel exponential increase in cost variability.

We will examine the relationship between comorbidity and health insurance costs and variability in costs among patients enrolled in health plans.

ELIGIBILITY:
Inclusion Criteria:

* patients with different burdens of comorbidity who have at least two continuous years of enrollment in the Generations Plus/ Northern Manhattan Health Network between June 2007 to July 2009 and members of a large self insured union trust fund from 2007-2010

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 15,000 patients who were continuously enrolled during the calendar years 2006 and 2010 in the Generations Plus/ Northern Manhattan Health Network and 226,000 members of a large self insured union trust fund from 2007-2010 will be combined. The data will include age, gender, length of plan enrollment, whether or not the patient is disabled, their diagnoses, and their use of medical and social services.
Sampling Method: Probability Sample
Enrollment: 241000 (Actual)
Dates: Start 2006-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Assessing costs & cost-variability among enrollees of health insurance programs utilizing Charlson's comorbidity index and administrative databases | The data within this dataset was collected between July 2006 and July 2010.
  Data for approximately 241,000 patients (15,000 who are members of the Generations Plus/ Northern Manhattan Health Network and 226,000 members of a large self insured union trust fund) during the calendar years 2006 and 2010 will be assembled and will include age, gender, length of plan enrollment, whether or not the patient is disabled, and their diagnoses. The data within this dataset was collected between July 2006 and July 2010.

CONTACTS AND LOCATIONS:
Locations (1):
- Generations Plus/ Northern Manhattan Health Network, The Bronx, New York, United States

REFERENCES:
- [Derived] Charlson M, Wells MT, Ullman R, King F, Shmukler C. The Charlson comorbidity index can be used prospectively to identify patients who will incur high future costs. PLoS One. 2014 Dec 3;9(12):e112479. doi: 10.1371/journal.pone.0112479. eCollection 2014. PMID 25469987